CLINICAL TRIAL: NCT02046239
Title: A Randomised Controlled Trial to Compare Subcuticular Suture vs Staples for Skin Closure After Liver Resection.
Brief Title: Suture vs Staples for Skin Closure After Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS13/10722
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Closure of the Skin After Liver Resection

ARMS (2):
- Staple Group (Other): Staple Group: At the end of the operation, the skin will be closed using stainless steel staples, which is standard clinical practice at St. James's University Hospital. Approximately ten days after the operation, the staples will be manually removed; this is normally performed by the patients GP.
  Interventions: Biological: Staple Group (control)
- Suture Group (Experimental): Suture Group: At the end of the operation, the skin will be closed using absorbable surgical suture. Manual removal of this suture is not required because the thread is self-absorbable.
  Interventions: Procedure: Suture Group

INTERVENTIONS:
Procedure: Suture Group
  Arms: Suture Group
Biological: Staple Group (control)
  Arms: Staple Group

SUMMARY:
Closure of the skin after liver resection (surgery to remove part of the liver) may be achieved by one of several methods. The standard method at our institution is to use stainless steel staples to adjoin the two sides of skin. Alternatively, a continuous absorbable suture may be used to "sew" the skin together.

The ideal method of closure should be safe, effective, associated with minimal patient discomfort and have a good cosmetic result. At present, there is no scientific evidence to describe which method is most suitable following liver resection.

The primary aims of this study is to investigate which method (subcuticular sutures vs staples) offers the best result in postoperative rate of (1) skin infection, (2) skin dehiscience (separation of skin) and (3) time taken to perform skin closure. In addition, we are interested in which method is best for patient satisfaction and cosmetic appearance and which method is most cost effective.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing liver resection surgery for benign or malignant aetiology
* All patients undergoing surgery as a living liver donor.

Exclusion Criteria:

* Any patient with an active wound infection
* Any patient with an active incisional wound hernia from previous surgery
* Synchronous bowel/liver surgery
* History of keloid formation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Post-operative infection time | 1 year

SECONDARY OUTCOMES:
Time taken for skin closure | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom